CLINICAL TRIAL: NCT03342235
Title: Excimer Laser Surgery for Anisometropic Amblyopia
Acronym: ATS19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not started due to lack of recruitment potential.
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS19; 2U10EY011751 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-11-14 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Anisometropic Amblyopia; Refractive Errors
Keywords: Excimer Laser Surgery; Photorefractive Keratectomy; Anisometropic Amblyopia; Visual Acuity; Refractive Surgical Procedures; PRK
MeSH Terms: conditions — Amblyopia; Refractive Errors | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Intervention Model Description: * Surgical Group: treatment with PRK and patching prescribed 2 hours per day with continued refractive correction (with spectacles and/or contact lenses) as able.
    o Surgery will be performed within 60 days of randomization
  * Non-surgical Control Group: patching prescribed 2 hours per day with continued refractive correction (with spectacles and/or contact lenses) as able.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Surgical Group (Experimental): Participants randomized to PRK surgery will be referred to a study surgical center. The participant will have a preoperative exam within 7 days prior to surgery and surgery within 60 days after randomization. Participants will continue prescribed 2 hours per day of patching between randomization and the day of surgery.
  Interventions: Procedure: Photorefractive Keratectomy (PRK); Device: Excimer Laser System
- Non-surgical Control Group (Active Comparator): For participants assigned to the non-surgical control group, patching will be prescribed for 2 hours per day with optical correction, and will continue until the 8-month primary outcome visit.
  Interventions: Other: Patching 2 hours per day

INTERVENTIONS:
Procedure: Photorefractive Keratectomy (PRK) — Subjects randomized to refractive surgery will be referred to one of six study surgical centers (surgical centers are listed in Appendix B) to have photorefractive keratectomy (PRK) in the affected eye within 60 days after randomization.
  Other Names: PRK Surgery
  Arms: Surgical Group
Other: Patching 2 hours per day — Patching prescribed 2 hours per day with continued refractive correction (with spectacles and/or contact lenses) as able.
  Other Names: Patching
  Arms: Non-surgical Control Group
Device: Excimer Laser System — Excimer Laser System for use in photorefractive keratectomy.
  Arms: Surgical Group

SUMMARY:
Study Objectives To compare the efficacy and safety of surgical treatment (PRK) versus non-surgical treatment of anisometropic amblyopia in children who have failed conventional treatment due to non-compliance or non-response.

Synopsis of Study Design

The study consists of two phases:

1. A Patching Run-In Phase during which all participants are treated for at least 8 weeks with continued refractive correction (with spectacles and/or contact lenses) and patching prescribed 42 hours per week (averaging 6 hours daily) until no further improvement over 2 consecutive visits at least 4 weeks apart or the vision no longer meets eligibility criteria.
2. A Randomized Trial Phase, beginning after no further VA improvement in the patching run-in phase and qualifying amblyopia is still present, during which the participant is assigned to either surgery with PRK and patching prescribed 2 hours per day or to non-surgical treatment with continued refractive correction (with spectacles and/or contact lenses) and patching prescribed 2 hours per day.

DETAILED DESCRIPTION:
The study is evaluating the efficacy of surgical treatment with PRK versus non-surgical treatment of anisometropic amblyopia in children who have failed conventional treatment. The primary analysis will be a treatment group comparison of the change in BCVA in the amblyopic eye at the 8-month primary outcome visit. For participants wearing a contact lens, the BCVA will be the visual acuity tested in the contact lens rather than in spectacles (or trial frames).

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to <8 years
2. Best-corrected amblyopic-eye VA using the ATS single-surround HOTV letter protocol (ATS-HOTV) meeting the following criteria:

   * If age 3 to <5 years, 20/80 to 20/800 (a re-test is required if the VA is 20/80)
   * If age 5 to <8 years, 20/63 to 20/800 (a re-test is required if the VA is 20/63)
   * Note: For participants who require a re-test (as specified above), the better of the test and re-test acuities must meet the eligibility criteria for the amblyopic eye and will serve as the enrollment VA.
3. Best-corrected fellow-eye VA meeting the following criteria by ATS-HOTV:

   * If age 3 years, 20/50 or better
   * If age 4 to 5 years, 20/40 or better
   * If age 6 to 7 years, 20/32 or better
4. Best-corrected inter-ocular acuity difference ≥ 3 logMAR lines by ATS-HOTV
5. Refractive error meeting the following criteria (based on a cycloplegic refraction that is not more than 4 months old):

   * Refractive error in the amblyopic eye must be greater than the fellow eye.
   * If the amblyopic eye is myopic, SE refractive error in the amblyopic eye between -3.00D and -12.00D, inclusive.
   * If the amblyopic eye is hyperopic, SE refractive error in the amblyopic eye between +3.00D and +6.00D, inclusive, if <=1.00D of astigmatism in the amblyopic eye; and between +3.00D and +5.00D, inclusive, if >1.00D of astigmatism in the amblyopic eye.
   * Astigmatism less than or equal to 3.50D in the amblyopic eye.
   * SE refractive error in the fellow eye between -4.00D and +3.00D, inclusive, with no astigmatism limits.
   * For participants 3 to <5 years of age, at least 5.00D of SE anisometropic difference between the two eyes by cycloplegic refraction; for subjects 5 to <8 years of age, at least 3.00D SE anisometropic difference
   * No more than 3.00D of difference in cylinder power between the two eyes
   * Target postoperative refractive error (if participant becomes eligible for randomization) must be achievable with PRK as defined in Table 3 and must be within 2.00D of the fellow eye.
6. Prior to enrollment into the Patching Run-In Phase, must have had patching and/or optical penalization with atropine or Bangerter filters prescribed for at least 6 months and optical correction of refractive error prescribed for at least 6 months. Prior treatment does not have to be continuous. Compliance with prescribed treatment does not influence eligibility but the best effort at compliance is expected from both the patient and provider.
7. Corneal thickness >500 microns (>510 microns within the previous 7 months, or corneal thickness between 500 and 510 microns within the last 2 months).
8. Central corneal thickness must be enough to allow the treatment dose needed while leaving a residual corneal thickness of ≥ 375 microns.
9. IOP ≤ 22 mm Hg within 7 months of enrollment
10. Investigator believes that the participant has achieved maximum improvement in amblyopic-eye VA with conventional treatment.
11. Investigator is willing to prescribe patching, and parent and child are willing to attempt patching for at least 8 weeks for 42 hours per week (averaging 6 hours daily) in the Patching Run-In Phase.
12. No rigid gas permeable lens (including OrthoK) worn in the past 2 months
13. Soft contact lens is currently worn, has been attempted within the past 4 months, or a contact lens fitting exam (paid for by the study) is scheduled or the investigator does the contact lens fitting on the same day as enrollment.
14. Parent understands the protocol and is willing to accept randomization (if child meets eligibility criteria after Patching Run-In Phase).
15. Parent has a phone (or access to phone) and is willing to be contacted by Jaeb Center staff or other study staff during the next 36 months.
16. Relocation outside of area of an active PEDIG site for this study without the next 36 months is not anticipated.

Exclusion Criteria:

1. Non-refractive ocular cause for reduced VA in the amblyopic eye (example: cataract, posterior staphyloma, extensive myelinated nerve fiber layer, optic nerve anomaly, macular scar, corneal opacity); or any cause of previous form deprivation.
2. Prior penetrating ocular surgery or injury
3. Prior strabismus surgery within 60 days preceding enrollment
4. Diagnosis of collagen vascular disease, Marfan syndrome, Ehlers-Danlos syndrome or other disorder of collagen synthesis
5. Previous ocular condition that may predispose the eye to be treated for future complications, for example:

   * Corneal disease (e.g., herpes simplex, herpes zoster keratitis, keratoconus or suspicion of keratoconus based upon family history, slit lamp exam, retinoscopy, or corneal topography (if able), recurrent erosion syndrome, corneal melt, or corneal dystrophy)
   * Established diagnosis of glaucoma
   * Any condition that, in the investigator's opinion, would interfere with or prolong corneal epithelial healing
   * History of significant eye rubbing or dry eye symptoms
6. History of retinopathy of prematurity resulting in macular ectopia
7. Down syndrome (trisomy 21)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity in the Amblyopic Eye | from randomization to the 8-month primary outcome visit
  Treatment group comparison of the change in Best-Corrected ATS-HOTV VA (BCVA) in the amblyopic eye at 8 months after randomization.
  ATS-HOTV = ATS single-surround HOTV testing protocol

SECONDARY OUTCOMES:
Randot Preschool Stereoacuity Outcomes by Treatment Group | At 8 months after randomization
  The distribution of Randot Preschool stereoacuity at randomization and the 8-month primary outcome visit will be tabulated separately for each treatment group. Change in stereoacuity from randomization to the 8-month visit will be tabulated for each group and compared between treatment groups using the exact Wilcoxon rank-sum test.
Refractive Error Outcomes in Surgery Group | At 7 months after randomization
  The distribution of change in refractive error in each eye at 7 months after randomization will be tabulated with computation of descriptive statistics. The difference between the 7-month refractive error and the target refractive error will be tabulated with computation of descriptive statistics.
Visual Acuity Outcomes | At 8 months
  A point estimate and corresponding 95% confidence interval will be calculated for the mean change in BCVA for the amblyopic-eye 8 months after baseline, adjusted for minimization covariates of age and VA at baseline as well as anisometropia type (hyperopia, myopia). The analyses will include data completed within the pre-specified analysis window for the 8-month visit after baseline and will follow a modified intent-to-treat principle as outlined for the primary analysis.
Distribution of refractive error outcomes | At 7 months after baseline
  The distribution of refractive error outcomes at 7 months after baseline will be tabulated with computation of descriptive statistics.
Distribution in Randot Preschool stereoacuity level | at baseline and 8 months
  The distribution in Randot Preschool stereoacuity level at baseline and 8 months after baseline and the change in stereoacuity for this interval will be tabulated and compared using a Wilcoxon signed rank test.
Visual Acuity Outcomes at 12 and 24 Months Post-surgery | at 12 and 24 months after surgery
  The distribution of the level and change in BCVA in the amblyopic eye at 12 and 24 months after surgery will be tabulated by treatment group with computation of descriptive statistics.
Stereoacuity at 12 and 24 Months Post-surgery | at 12 and 24 months after surgery
  The distribution of Randot Preschool stereoacuity and change in stereoacuity at the 12- and 24-month post-surgery visits will be tabulated separately for each treatment group
Refractive Error at 12 and 24 Months Post-surgery | at 12 and 24 months after surgery
  The distribution of change in refractive error in each eye at 12 and 24 months after surgery will be tabulated by treatment group with computation of descriptive statistics. The difference between the refractive errors at these visits and the target refractive error will be tabulated by treatment group with computation of descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn A Paysse, MD, Study Chair — Baylor College of Medicine; David K Wallace, MD, MPH, Study Chair — Duke Eye Center

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.
URL: http://pedig.net